CLINICAL TRIAL: NCT02302898
Title: Characteristics Associated With Weight Regain After Roux-en-Y Gastric Bypass
Brief Title: Roux-en-Y Gastric Bypass and Weight Regain
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201409107
Record Dates: First submitted 2014-11-19; First posted 2014-11-27 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Obesity
Keywords: Roux-en-Y Gastric Bypass Surgery; Weight Regain
MeSH Terms: conditions — Obesity | interventions — National Cancer Institute (U.S.)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Wt maintenance: Eating Behavior Evaluation Measurement of Functional gastric volume Measurement of gastric pouch and GJ sizes
  Interventions: Behavioral: Eating Behavior Evaluation; Other: Measurement of Functional gastric volume; Other: Measurement of gastric pouch and GJ size
- Wt Regain: Eating Behavior Evaluation Measurement of Functional gastric volume Measurement of gastric pouch and GJ sizes
  Interventions: Behavioral: Eating Behavior Evaluation; Other: Measurement of Functional gastric volume; Other: Measurement of gastric pouch and GJ size

INTERVENTIONS:
Behavioral: Eating Behavior Evaluation — Scores will be measured on binge eating behaviors and an increased craving for sweets.
  Other Names: Yale Food Addiction Scale (YFAS); Eating Disorder Examination (EDE); The Food Craving Inventory (FCI); National Cancer Institute (NCI) ASA24
Other: Measurement of Functional gastric volume — The functional gastric volume is the amount of food or liquid that can be consumed to a feeling of comfortably full in one meal.
Other: Measurement of gastric pouch and GJ size — Anatomical dimensions of the gastric pouch and GJ will be determined by using an articulated measuring tool during upper GI tract endoscopy.

SUMMARY:
This study compares eating behaviors, meal size, and the size of the gastric pouch and connection between the gastric pouch and small intestine in patients who had gastric bypass surgery two or more years ago and regained weight compared with patients who had gastric bypass surgery two or more years ago and maintained their weight loss.

DETAILED DESCRIPTION:
Obesity affects a third of adults in the United States. The most effective treatment for weight loss is bariatric surgery, and the most common surgery performed in the US is Roux-en-Y Gastric Bypass (RYGB). However, a significant number of patients regain weight that was lost after surgery. The mechanisms for weight regain are likely multifactorial, but not well understood. Disordered eating behaviors and dilated gastrojejunostomies (GJ), which presumably allows a patient to consume larger portion sizes during a meal, correlate with weight regain. Moreover, some data suggest that changes to the gut anatomy may drive eating behaviors and food preferences. However, no studies have simultaneously evaluated functional gastric volume (the volume of solid or liquid food that can be consumed to a level of comfortable fullness in one sitting), anatomical gastric pouch size and GJ diameter, and eating behaviors in patients who maintained their post RYGB weight compared with patients who have regained weight from their maximum weight loss after RYGB to determine the relationship among post RYGB eating behavior, functional and anatomical gastric pouch size, GJ diameter and weight change. Accordingly, the objectives of this proposal are to compare 1) eating behaviors 2) functional gastric volume and 3) anatomical dimensions of the gastric pouch and GJ in patients who are >2 years post RYGB and have regained >20% of their maximum lost weight and those who are >2 years post RYGB and have maintained at least 90% weight loss since surgery. The following specific aims will be evaluated:

Aim 1. Evaluate whether differences in eating behaviors exist between subjects who have maintained weight loss after RYGB or regained >20% of their maximum lost weight. The investigators hypothesize that subjects who have regained weight after RYGB will have higher scores on binge eating behaviors and an increased craving for sweets compared with patients who have maintained weight loss after RYGB. Eating behaviors will be determined by performing the Yale Food Addiction Scale (YFAS), Eating Disorder Examination (EDE), The Food Craving Inventory (FCI), and the National Cancer Institute (NCI) ASA24.

Aim 2. Evaluate whether differences exist in functional gastric volume between subjects who have maintained weight loss after RYGB or regained >20% of their maximum lost weight. The investigators hypothesize that patients who have regained weight after RYGB will have an increased functional gastric volume to both solids and liquids compared to subjects who have maintained weight loss after RYGB. Functional gastric volume will be measured during both a solid and liquid meal test.

Aim 3. Evaluate whether differences exist in gastric pouch and GJ sizes between subjects who have maintained weight loss after RYGB or regained >20% of their maximum lost weight. The investigators hypothesize that patients who have regained weight after RYGB will have increased gastric pouch size and GJ diameter compared with patients who have maintained their weight loss after RYGB. Anatomical dimensions of the gastric pouch and GJ will be determined by using an articulated measuring tool during upper GI tract endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Ages of 21 and 60
* Laparoscopic RYGB surgery >2 years before screening
* Regained >20% weight from their maximum weight lost after surgery or maintained at least 90% weight loss from the maximum weight loss after surgery

Exclusion Criteria:

* Allergy to lidocaine, nut allergies, milk intolerance or any other food allergies/restrictions that are included in our test meals
* A history of alcohol abuse
* Currently consuming >20 gm of alcohol per day
* Greater than 2 points on the MAST
* Severe organ dysfunction
* Anemia (hemoglobin <10mg/dl)
* PT, PTT and INR > 1.5x UNL
* Triglycerides > 400
* LFT > 2x UNL
* Women who are pregnant or lactating
* Participants that smoke greater than 20 pack years
* Actively using illegal drugs
* Depression or other psychological disorders that are untreated
* Diabetics receiving Insulin
* Patients that have been hospitalized and/or had surgery in the last three months that may be unstable (PI will determine this at Physical Exam)

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will consist of 20 patients who had laparoscopic RYGB surgery >2 years before screening and have regained >20% weight from their maximum weight lost after surgery and 20 patients who had laparoscopic RYGB surgery >2 years before screening and have maintained at least 90% weight loss from the maximum weight loss after surgery. These patients will be identified from the bariatric surgical population at Washington University School of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2015-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Eating Behavior Assessment scores will be compared between both groups | Greater than 2 years post RYGB
  Eating behaviors will be determined by performing the Yale Food Addiction Scale (YFAS), Eating Disorder Examination (EDE), The Food Craving Inventory (FCI), and the National Cancer Institute (NCI) ASA24.

SECONDARY OUTCOMES:
Functional gastric volume will be measured | Greater than 2 years post RYGB
  The functional gastric volume is the amount of food or liquid that can be consumed to a feeling of comfortably full in one meal.
Gastric pouch size and GJ diameter will be measured | Greater than 2 years post RYGB
  Anatomical dimensions of the gastric pouch and GJ will be determined by using an articulated measuring tool during upper GI tract endoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Shelby Sullivan, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Pories WJ, Swanson MS, MacDonald KG, Long SB, Morris PG, Brown BM, Barakat HA, deRamon RA, Israel G, Dolezal JM, et al. Who would have thought it? An operation proves to be the most effective therapy for adult-onset diabetes mellitus. Ann Surg. 1995 Sep;222(3):339-50; discussion 350-2. doi: 10.1097/00000658-199509000-00011. PMID 7677463
- [Background] Magro DO, Geloneze B, Delfini R, Pareja BC, Callejas F, Pareja JC. Long-term weight regain after gastric bypass: a 5-year prospective study. Obes Surg. 2008 Jun;18(6):648-51. doi: 10.1007/s11695-007-9265-1. Epub 2008 Apr 8. PMID 18392907
- [Background] Brethauer SA, Aminian A, Romero-Talamas H, Batayyah E, Mackey J, Kennedy L, Kashyap SR, Kirwan JP, Rogula T, Kroh M, Chand B, Schauer PR. Can diabetes be surgically cured? Long-term metabolic effects of bariatric surgery in obese patients with type 2 diabetes mellitus. Ann Surg. 2013 Oct;258(4):628-36; discussion 636-7. doi: 10.1097/SLA.0b013e3182a5034b. PMID 24018646
- [Background] Freire RH, Borges MC, Alvarez-Leite JI, Toulson Davisson Correia MI. Food quality, physical activity, and nutritional follow-up as determinant of weight regain after Roux-en-Y gastric bypass. Nutrition. 2012 Jan;28(1):53-8. doi: 10.1016/j.nut.2011.01.011. Epub 2011 Aug 31. PMID 21885246
- [Background] Schultes B, Ernst B, Wilms B, Thurnheer M, Hallschmid M. Hedonic hunger is increased in severely obese patients and is reduced after gastric bypass surgery. Am J Clin Nutr. 2010 Aug;92(2):277-83. doi: 10.3945/ajcn.2009.29007. Epub 2010 Jun 2. PMID 20519559
- [Background] Miras AD, Jackson RN, Jackson SN, Goldstone AP, Olbers T, Hackenberg T, Spector AC, le Roux CW. Gastric bypass surgery for obesity decreases the reward value of a sweet-fat stimulus as assessed in a progressive ratio task. Am J Clin Nutr. 2012 Sep;96(3):467-73. doi: 10.3945/ajcn.112.036921. Epub 2012 Jul 25. PMID 22836034
- [Background] Pepino MY, Bradley D, Eagon JC, Sullivan S, Abumrad NA, Klein S. Changes in taste perception and eating behavior after bariatric surgery-induced weight loss in women. Obesity (Silver Spring). 2014 May;22(5):E13-20. doi: 10.1002/oby.20649. Epub 2013 Dec 6. PMID 24167016
- [Background] Hsu LK, Betancourt S, Sullivan SP. Eating disturbances before and after vertical banded gastroplasty: a pilot study. Int J Eat Disord. 1996 Jan;19(1):23-34. doi: 10.1002/(SICI)1098-108X(199601)19:13.0.CO;2-Y. PMID 8640199
- [Background] White MA, Kalarchian MA, Masheb RM, Marcus MD, Grilo CM. Loss of control over eating predicts outcomes in bariatric surgery patients: a prospective, 24-month follow-up study. J Clin Psychiatry. 2010 Feb;71(2):175-84. doi: 10.4088/JCP.08m04328blu. Epub 2009 Oct 20. PMID 19852902
- [Background] Saunders R. "Grazing": a high-risk behavior. Obes Surg. 2004 Jan;14(1):98-102. doi: 10.1381/096089204772787374. PMID 14980042
- [Result] Christou NV, Look D, Maclean LD. Weight gain after short- and long-limb gastric bypass in patients followed for longer than 10 years. Ann Surg. 2006 Nov;244(5):734-40. doi: 10.1097/01.sla.0000217592.04061.d5. PMID 17060766
- [Result] Sjostrom L, Lindroos AK, Peltonen M, Torgerson J, Bouchard C, Carlsson B, Dahlgren S, Larsson B, Narbro K, Sjostrom CD, Sullivan M, Wedel H; Swedish Obese Subjects Study Scientific Group. Lifestyle, diabetes, and cardiovascular risk factors 10 years after bariatric surgery. N Engl J Med. 2004 Dec 23;351(26):2683-93. doi: 10.1056/NEJMoa035622. PMID 15616203
- [Result] Franco JV, Ruiz PA, Palermo M, Gagner M. A review of studies comparing three laparoscopic procedures in bariatric surgery: sleeve gastrectomy, Roux-en-Y gastric bypass and adjustable gastric banding. Obes Surg. 2011 Sep;21(9):1458-68. doi: 10.1007/s11695-011-0390-5. PMID 21455833
- [Result] Buchwald H, Avidor Y, Braunwald E, Jensen MD, Pories W, Fahrbach K, Schoelles K. Bariatric surgery: a systematic review and meta-analysis. JAMA. 2004 Oct 13;292(14):1724-37. doi: 10.1001/jama.292.14.1724. PMID 15479938
- [Result] Hall JC, Watts JM, O'Brien PE, Dunstan RE, Walsh JF, Slavotinek AH, Elmslie RG. Gastric surgery for morbid obesity. The Adelaide Study. Ann Surg. 1990 Apr;211(4):419-27. doi: 10.1097/00000658-199004000-00007. PMID 2181950
- [Result] Ullrich J, Ernst B, Wilms B, Thurnheer M, Schultes B. Roux-en Y gastric bypass surgery reduces hedonic hunger and improves dietary habits in severely obese subjects. Obes Surg. 2013 Jan;23(1):50-5. doi: 10.1007/s11695-012-0754-5. PMID 22941334
- [Result] Hsu LK, Benotti PN, Dwyer J, Roberts SB, Saltzman E, Shikora S, Rolls BJ, Rand W. Nonsurgical factors that influence the outcome of bariatric surgery: a review. Psychosom Med. 1998 May-Jun;60(3):338-46. doi: 10.1097/00006842-199805000-00021. PMID 9625222
- [Result] Kalarchian MA, Marcus MD, Wilson GT, Labouvie EW, Brolin RE, LaMarca LB. Binge eating among gastric bypass patients at long-term follow-up. Obes Surg. 2002 Apr;12(2):270-5. doi: 10.1381/096089202762552494. PMID 11975227
- [Result] Kofman MD, Lent MR, Swencionis C. Maladaptive eating patterns, quality of life, and weight outcomes following gastric bypass: results of an Internet survey. Obesity (Silver Spring). 2010 Oct;18(10):1938-43. doi: 10.1038/oby.2010.27. Epub 2010 Feb 18. PMID 20168309
- [Result] Livhits M, Mercado C, Yermilov I, Parikh JA, Dutson E, Mehran A, Ko CY, Gibbons MM. Preoperative predictors of weight loss following bariatric surgery: systematic review. Obes Surg. 2012 Jan;22(1):70-89. doi: 10.1007/s11695-011-0472-4. PMID 21833817
- [Result] Cooper Z, Cooper PJ, Fairburn CG. The validity of the eating disorder examination and its subscales. Br J Psychiatry. 1989 Jun;154:807-12. doi: 10.1192/bjp.154.6.807. PMID 2597887
- [Result] Fairburn CG, Cooper Z. Binge eating: Nature, assessment and treatment. In: Fairburn CG, Wilson G, eds. The Eating Disorder Examination. 12 ed. New York, New York: Guilford Press, 1993:317-360.
- [Result] White MA, Whisenhunt BL, Williamson DA, Greenway FL, Netemeyer RG. Development and validation of the food-craving inventory. Obes Res. 2002 Feb;10(2):107-14. doi: 10.1038/oby.2002.17. PMID 11836456
- [Result] Gearhardt AN, Corbin WR, Brownell KD. Preliminary validation of the Yale Food Addiction Scale. Appetite. 2009 Apr;52(2):430-6. doi: 10.1016/j.appet.2008.12.003. Epub 2008 Dec 11. PMID 19121351
- [Result] Subar AF, Kirkpatrick SI, Mittl B, Zimmerman TP, Thompson FE, Bingley C, Willis G, Islam NG, Baranowski T, McNutt S, Potischman N. The Automated Self-Administered 24-hour dietary recall (ASA24): a resource for researchers, clinicians, and educators from the National Cancer Institute. J Acad Nutr Diet. 2012 Aug;112(8):1134-7. doi: 10.1016/j.jand.2012.04.016. Epub 2012 Jun 15. No abstract available. PMID 22704899
- [Result] Flanagan L. Measurement of Functional Pouch Volume following the Gastric Bypass Procedure. Obes Surg. 1996 Feb;6(1):38-43. doi: 10.1381/096089296765557240. PMID 10731248
- [Result] Laurenius A, Larsson I, Bueter M, Melanson KJ, Bosaeus I, Forslund HB, Lonroth H, Fandriks L, Olbers T. Changes in eating behaviour and meal pattern following Roux-en-Y gastric bypass. Int J Obes (Lond). 2012 Mar;36(3):348-55. doi: 10.1038/ijo.2011.217. Epub 2011 Nov 29. PMID 22124454
- [Result] Abu Dayyeh BK, Lautz DB, Thompson CC. Gastrojejunal stoma diameter predicts weight regain after Roux-en-Y gastric bypass. Clin Gastroenterol Hepatol. 2011 Mar;9(3):228-33. doi: 10.1016/j.cgh.2010.11.004. Epub 2010 Nov 17. PMID 21092760
- [Result] Heneghan HM, Yimcharoen P, Brethauer SA, Kroh M, Chand B. Influence of pouch and stoma size on weight loss after gastric bypass. Surg Obes Relat Dis. 2012 Jul-Aug;8(4):408-15. doi: 10.1016/j.soard.2011.09.010. Epub 2011 Sep 23. PMID 22055390
- [Result] Hallowell PT, Stellato TA, Yao DA, Robinson A, Schuster MM, Graf KN. Should bariatric revisional surgery be avoided secondary to increased morbidity and mortality? Am J Surg. 2009 Mar;197(3):391-6. doi: 10.1016/j.amjsurg.2008.11.011. PMID 19245921
- [Result] Zingg U, McQuinn A, DiValentino D, Kinsey-Trotman S, Game P, Watson D. Revisional vs. primary Roux-en-Y gastric bypass--a case-matched analysis: less weight loss in revisions. Obes Surg. 2010 Dec;20(12):1627-32. doi: 10.1007/s11695-010-0214-z. PMID 20577830
- [Result] Radtka JF 3rd, Puleo FJ, Wang L, Cooney RN. Revisional bariatric surgery: who, what, where, and when? Surg Obes Relat Dis. 2010 Nov-Dec;6(6):635-42. doi: 10.1016/j.soard.2010.04.005. Epub 2010 May 4. PMID 20702147
- [Result] Morales MP, Wheeler AA, Ramaswamy A, Scott JS, de la Torre RA. Laparoscopic revisional surgery after Roux-en-Y gastric bypass and sleeve gastrectomy. Surg Obes Relat Dis. 2010 Sep-Oct;6(5):485-90. doi: 10.1016/j.soard.2009.09.022. Epub 2010 Jan 1. PMID 20870181
- [Result] Thompson CC, Slattery J, Bundga ME, Lautz DB. Peroral endoscopic reduction of dilated gastrojejunal anastomosis after Roux-en-Y gastric bypass: a possible new option for patients with weight regain. Surg Endosc. 2006 Nov;20(11):1744-8. doi: 10.1007/s00464-006-0045-0. Epub 2006 Oct 5. PMID 17024527
- [Result] Herron DM, Birkett DH, Thompson CC, Bessler M, Swanstrom LL. Gastric bypass pouch and stoma reduction using a transoral endoscopic anchor placement system: a feasibility study. Surg Endosc. 2008 Apr;22(4):1093-9. doi: 10.1007/s00464-007-9623-z. Epub 2007 Nov 20. PMID 18027049
- [Result] Thompson CC, Chand B, Chen YK, DeMarco DC, Miller L, Schweitzer M, Rothstein RI, Lautz DB, Slattery J, Ryan MB, Brethauer S, Schauer P, Mitchell MC, Starpoli A, Haber GB, Catalano MF, Edmundowicz S, Fagnant AM, Kaplan LM, Roslin MS. Endoscopic suturing for transoral outlet reduction increases weight loss after Roux-en-Y gastric bypass surgery. Gastroenterology. 2013 Jul;145(1):129-137.e3. doi: 10.1053/j.gastro.2013.04.002. Epub 2013 Apr 5. PMID 23567348
- [Result] Thompson CC, Jacobsen GR, Schroder GL, Horgan S. Stoma size critical to 12-month outcomes in endoscopic suturing for gastric bypass repair. Surg Obes Relat Dis. 2012 May-Jun;8(3):282-7. doi: 10.1016/j.soard.2011.03.014. Epub 2011 Apr 19. PMID 21640665
- [Result] Jirapinyo P, Slattery J, Ryan MB, Abu Dayyeh BK, Lautz DB, Thompson CC. Evaluation of an endoscopic suturing device for transoral outlet reduction in patients with weight regain following Roux-en-Y gastric bypass. Endoscopy. 2013 Jul;45(7):532-6. doi: 10.1055/s-0032-1326638. Epub 2013 Jun 25. PMID 23801313
- [Result] Abu Dayyeh BK, Ryan MB, Thompson CC. 309 Ghrelin and Gastric Pouch Parameters Are Associated With Feeding Behaviors After Roux-en-Y Gastric Bypass. Gastroenterology 2013;144:S-64.
- [Result] Selzer ML. The Michigan alcoholism screening test: the quest for a new diagnostic instrument. Am J Psychiatry. 1971 Jun;127(12):1653-8. doi: 10.1176/ajp.127.12.1653. No abstract available. PMID 5565851
- [Result] Geliebter A, Gibson CD, Hernandez DB, Atalayer D, Kwon A, Lee MI, Mehta N, Phair D, Gluck ME. Plasma cortisol levels in response to a cold pressor test did not predict appetite or ad libitum test meal intake in obese women. Appetite. 2012 Dec;59(3):956-9. doi: 10.1016/j.appet.2012.08.025. Epub 2012 Sep 13. PMID 22983369
- [Result] Sullivan S, Stein R, Jonnalagadda S, Mullady D, Edmundowicz S. Aspiration therapy leads to weight loss in obese subjects: a pilot study. Gastroenterology. 2013 Dec;145(6):1245-52.e1-5. doi: 10.1053/j.gastro.2013.08.056. Epub 2013 Sep 6. PMID 24012983